CLINICAL TRIAL: NCT00001554
Title: Intraoperative Infrared Functional Brain Mapping
Brief Title: Infrared Camera for Brain Mapping During Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 960093; 96-N-0093
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-05

CONDITIONS: Epilepsy; Neurologic Manifestations
Keywords: Cortical Localization; Optical Imaging; Thermal Imaging
MeSH Terms: conditions — Epilepsy; Neurologic Manifestations | interventions — Neuroimaging

INTERVENTIONS:
Device: intraoperative infrared (IR) neuroimaging

SUMMARY:
It is extremely important to identify and distinguish healthy brain tissue from diseased brain tissue during neurosurgery. If normal tissue is damaged during neurosurgery it can result in long term neurological problems for the patient.

The brain tissue as it appears prior to the operation on CT scan and MRI is occasionally very different from how it appears during the actual operation. Therefore, it is necessary to develop diagnostic procedures that can be used during the operation

Presently, the techniques used for intraoperative mapping of the brain are not reliable in all cases in which they are used. Researchers in this study have developed a new approach that may allow diseased brain tissue to be located during an operation with little risk. This new approach uses nfrared technology to locate the diseased tissue and identify healthy brain tissue.

The goal of this study is to investigate the clinical use of intraoperative infrared (IR) neuroimaging to locate diseased tissue and distinguish it from normal functioning tissue during the operation.

DETAILED DESCRIPTION:
It is important during neurosurgical procedures to identify and preserve eloquent functional cortex adjacent to a resectable lesion. Resection of a lesion infiltrating vital cerebral cortex can be associated with postoperative neurological deficits if the surgeon cannot clearly distinguish between the infiltrating borders of a lesion and surrounding functionally eloquent tissue. Spatial relationships between a lesion and surrounding normal brain can change significantly from those determined by preoperative methods such as CT and MRI scans. Necessary intraoperative interventions such as cerebrospinal fluid drainage, osmotic diuresis and lesion debulking cause quantitatively unpredictable brain shift in three dimensions. Therefore functional localization in real time that can be performed in the operating room is desirable. However, intraoperative real-time functional mapping techniques now available cannot be used in many surgical situations and are not sufficiently reliable in all cases in which they are used.

We have developed an intraoperative approach that may permit reliable lesion localization and brain functional mapping in real time with minimal risk. This approach makes use of infrared technology to identify functionally active eloquent cortex and may differentiate abnormal tissue from normal cortex.

The goal of this study is to investigate the clinical use of intraoperative infrared (IR) neuroimaging to differentiate intracranial lesions from surrounding normal functionally important tissue in real time. Reliable real-time intraoperative functional mapping of eloquent cortex adjacent to lesions by this technique would improve the safety and effectiveness of many neurosurgical procedures.

ELIGIBILITY:
Adult patients who will be undergoing craniotomy for lesions such as tumor, epileptic focus, vascular malformation or infection.

Adult patients who are able to provide informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80
Dates: Start 1996-06; Study Completion 2000-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Brugge JF, Poon PW, So AT, Wu BM, Chan FH, Lam FK. Thermal images of somatic sensory cortex obtained through the skull of rat and gerbil. Exp Brain Res. 1995;106(1):7-18. doi: 10.1007/BF00241352. PMID 8542979
- [Background] George JS, Lewine JD, Goggin AS, Dyer RB, Flynn ER. IR thermal imaging of a monkey's head: local temperature changes in response to somatosensory stimulation. Adv Exp Med Biol. 1993;333:125-36. doi: 10.1007/978-1-4899-2468-1_12. No abstract available. PMID 8362657